CLINICAL TRIAL: NCT03232008
Title: The Effects of Canderel (Aspartame and Acesulfame-k Blend) on Blood Glucose Concentration and Appetite Scores in Humans: a Randomised Controlled Trial
Brief Title: Canderel:Effects on Blood Glucose Concentration and Appetite Scores
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Dr Christopher Corpe, Nutrition Sciences Lecturer, Principal investigator, King's College London
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: KCLMScNutr2017
Record Dates: First submitted 2017-06-19; First posted 2017-07-27 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Appetitive Behavior; Glucose Metabolism Disorders
Keywords: Blood glucose; Appetite
MeSH Terms: conditions — Appetitive Behavior; Glucose Metabolism Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Experiment A- experimental (Experimental): 3g Canderel in 250ml water
  Interventions: Dietary Supplement: Canderel drink
- Experiment A- control (No Intervention): 3g of maltodextrin in 250 ml of water
- Experiment B- experimental (Experimental): 3g Canderel + 35g Lyle's Golden Syrup in 250 ml water
  Interventions: Dietary Supplement: Canderel+Lyle's Golden Syrup drink
- Experiment B- control (No Intervention): 3g Lyle's Golden Syrup + 35g of maltodextrin in 250 ml of water

INTERVENTIONS:
Dietary Supplement: Canderel drink — 1.4% aspartame and 0.95% acesulfame-k and 95% maltodextrin; 3g dissolved in 250ml of water
  Arms: Experiment A- experimental
Dietary Supplement: Canderel+Lyle's Golden Syrup drink — Canderel: 1.4% aspartame and 0.95% acesulfame-k and 95% maltodextrin; 3g dissolved in 250ml of water Lyle's Golden Syrup: 35 g (27g of glucose and fructose)
  Arms: Experiment B- experimental

SUMMARY:
This study investigates the effects of Canderel, an aspartame and acesulfame-k blend artificial sweetener powder, on post-postprandial blood glucose levels and appetite scores.

DETAILED DESCRIPTION:
The study is separated into two parts: A) investigating the effects of artificial sweeteners in combination with complex carbohydrates; and B) investigating the effects of artificial sweeteners in combination with simple sugars.

A) Participants will be randomly given either the placebo drink (3g of maltodextrin dissolved in 250ml of water) or the Canderel drink (3g of Canderel dissolved in 250ml of water) alongside an isocaloric high carbohydrate breakfast. Blood glucose measurements will be obtained through finger pricking and appetite will be measured using self-reported visual analog scores rating hunger, desire to eat, fullness and alertness for up to 3 hours after breakfast.

B)Participants will be randomly given either the placebo drink (3g of Lyle's Golden syrup and 3g of maltodextrin dissolved in 250ml of water) or the Canderel+sugars drink (3g of Canderel and 3g of Lyle's Golden syrup dissolved in 250ml of water) . Blood glucose measurements will be obtained through finger pricking and appetite will be measured using self-reported visual analog scores rating hunger, desire to eat, fullness and alertness for up to 3 hours after drink

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults (18-64)

Exclusion Criteria:

-

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2021-03-28 (Estimated)

PRIMARY OUTCOMES:
Change in Blood glucose | 0-180min (Measured from baseline to 90min every 15min; 90-180min every 30min)
  Capillary blood obtained from fingerprick and measured using glucose monitor
Change in Appetite | 0-180min (Measured from baseline to 90min every 15min; 90-180min every 30min)
  Feelings of hunger, desire to eat, fullness and alertness measured using Visual Analog Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Christopher Corpe, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No